CLINICAL TRIAL: NCT02616822
Title: Acute Effects Of Trans-Resveratrol in Endothelial Function in Treated Hypertensive Patients
Brief Title: Effects of Trans-Resveratrol in Endothelial Function in Hypertensive Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hospital Universitario Pedro Ernesto (Other)
Responsible Party: Principal Investigator, Bianca Cristina Antunes Alves Marques, RD, Master student, Hospital Universitario Pedro Ernesto
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Resv2013
Record Dates: First submitted 2015-10-16; First posted 2015-11-30 (Estimated); Last update posted 2015-11-30 (Estimated); Status verified 2015-11

CONDITIONS: Endothelial Dysfunction
Keywords: hypertension; endothelium; resveratrol; clinical trials
MeSH Terms: conditions — Hypertension | interventions — Resveratrol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- trans-resveratrol (Experimental): Used for trans-resveratrol substance 300 mg single dose
  Interventions: Dietary Supplement: Trans-resveratrol
- Placebo (Placebo Comparator): Used for placebo substance single dose
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Trans-resveratrol — Used for trans-resveratrol substance 300 mg single dose
  Arms: trans-resveratrol
Other: Placebo — Used for placebo substance single dose
  Arms: Placebo

SUMMARY:
Arterial Hypertension (HBP) has a high prevalence and low rates of control, is considered a major modifiable risk factors and one of the most important public health problems. Mortality from cardiovascular disease increases progressively with increasing blood pressure (BP) in a linear, continuous and independent. The pathophysiological mechanisms involved in the pathogenesis of hypertension exhibit metabolic abnormalities, which are related to endothelial dysfunction. Resveratrol, a polyphenol stilbene derived from various species of plants, but in our food, mainly present in red wine and grapes, has shown protective effects in cardiovascular diseases, such as preventing the damage caused by oxidative stress, decreased plasma lipids with inhibiting the formation of atherosclerotic plaque; protective effect of vascular endothelium, with increased release of nitric oxide and decreased production of free radicals in animal models, but human studies are limited and insufficient to clarify the possible effects of trans-resveratrol (biologically active form) on endothelial function, blood pressure and central aortic pressure in treated hypertensive individuals.The aim of this study is to evaluate the acute effects of trans-resveratrol supplementation on endothelial function in treated hypertensive patients.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients aged between 45 and 65 years, of both genders.
* Patients with a previous diagnosis of hypertension.
* Patients with endothelial disfunction.
* Stable use of antihypertensive treatment for at least 2 months.
* Patients with food consumption maintained for at least 4 weeks, oriented to limit the intake of foods rich in polyphenols, such as peanut butter, cranberry, blackberry, red grapes, red wine, green tea and chocolate.
* Signing the consent form.

Exclusion Criteria:

* Smoking.
* Diabetes Mellitus and / or use of insulin or oral hypoglycemic agents.
* Hormone replacement therapy.
* Use of ß-blockers and statins.
* Sleep apnea.
* Changes in thyroid function, chronic renal and liver diseases.
* Clinically evident coronary heart disease with previous myocardial infarction and / or revascularization, with clinical signs of heart failure, cardiac arrhythmia, symptomatic or clinically significant valvular disease, prior stroke.
* History of drug or alcohol abuse. Presence of some kind of eating disorder;
* Diets restricted by choice (vegetarianism, carbohydrate restriction);
* Use of nutritional supplements (vitamins, minerals), to at least seven (7) days prior to the study;
* Patients who have any severe illness and life-threatening any condition, disease or therapy that, in the opinion of the investigator, may adversely affect the results, interfere with the study objectives or jeopardize the safety of patients.

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-01; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Flow-mediated dilatation of the brachial artery | 90 minutes
  The patient lay comfortably in the supine position with slightly abducted right arm. After located the brachial artery, the transducer was placed on the anteromedial face of the right arm, perpendicular to the axis of the arm, 5-10 cm above the antecubital crease on the artery. The basal diameter of the brachial artery (BBAD) and post occlusion brachial artery diameter (POBAD) were measured manually between the intima-lumen interfaces at end-diastole. After BBAD, the site of contact of the probe was marked on the skin, so that the measurement of POBAD occur at the same site. The occlusion is maintained for five minutes through cuff on the arm, which print pressure slightly above the systolic blood pressure, confirmed by no pulse Doppler. The POBAD was measured 30, 60 and 90 seconds after releasing the flow. At baseline, after checking the criteria for inclusion and exclusion and signing the informed consent, the selected patient performs the DMF fasting and after 90 minutes.

SECONDARY OUTCOMES:
Determination of central aortic pressure (Sphygmocor) | 90 minutes
  Noninvasive test, conducted in peaceful environment, temperature controlled, patient lying supine, using his right arm to measure blood pressure and central aortic pressure.
  The analysis of radial artery pulse wave by applanation tonometry is performed to derive central artery pressures and other hemodynamic parameters using Sphygmocor system (Atcor, USA). After measuring the BP in the brachial artery pulse wave of the radial artery on the same side were obtained for at least 10 seconds using a tonometer (SPC-301 - Millar Instruments, Houston, Texas), calibrated according to the brachial BP. The resulting radial pulse waves are processed using specific software (Sphygmocor v7 AtCor, USA) to derive the corresponding central aortic pressure through a previously validated transfer function. At baseline, after checking the criteria for inclusion and exclusion and signing the informed consent, the selected patient performs the SphymoCor fasting and after 90 minutes.